CLINICAL TRIAL: NCT01908868
Title: A Trial of EBUS-TBNA Versus Conventional TBNA in Diagnosis of Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1Trg/PG-2012/12563-601
Record Dates: First submitted 2013-07-16; First posted 2013-07-26 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EBUS-TBNA (Experimental): EBUS-TBNA (with endobronchial and transbronchial lung biopsy)
  Interventions: Other: EBUS-TBNA; Other: Endobronchial and transbronchial biopsy
- Conventional TBNA (Active Comparator): Conventional TBNA (with endobronchial and transbronchial lung biopsy)
  Interventions: Other: Conventional TBNA; Other: Endobronchial and transbronchial biopsy

INTERVENTIONS:
Other: EBUS-TBNA — Mediastinal and hilar lymph node aspiration using endobronchial ultrasound
  Arms: EBUS-TBNA
Other: Conventional TBNA — Mediastinal and hilar lymph node aspiration using blind transbronchial needle aspiration
  Arms: Conventional TBNA
Other: Endobronchial and transbronchial biopsy — Endobronchial and transbronchial lung biopsy using flexible bronchoscopy

SUMMARY:
The investigators hypothesize that conventional or EBUS-TBNA will have equal efficiency in diagnosing sarcoidosis when performed in conjunction with endobronchial and transbronchial lung biopsy.

DETAILED DESCRIPTION:
Diagnostic procedures like transbronchial lung biopsy (TBLB), transbronchial needle aspiration (TBNA) and endobronchial biopsy (EBB) are routinely used to obtain pathological confirmation of pulmonary sarcoidosis. Real-time convex probe endobronchial ultrasound-guided TBNA (EBUS-TBNA) has shown immense potential, however it is costly, labor intensive and still has limited availability, especially in low and middle income countries. In the past, TBLB has been the bronchoscopic procedure of choice for diagnosis of sarcoidosis however currently its role is being debated with the advent of EBUS. We have observed that EBUS even though has high yield yet the optimal diagnosis is obtained only when combined with EBB and TBLB. The investigators hypothesize that conventional or EBUS-TBNA will have equal efficiency in diagnosing sarcoidosis when performed in conjunction with endobronchial and transbronchial lung biopsy.

The study compares the diagnostic yield of EBUS-TBNA (plus EBB and TBLB) vs. conventional TBNA (plus EBB and TBLB) for diagnosis of sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients presenting with clinicoradiological features suggestive of sarcoidosis and an indication for transbronchial needle aspiration

Exclusion Criteria:

* Pregnancy
* Hypoxemia (SpO2 <90%) on room air
* Poor lung function (forced expiratory volume in first second [FEV1] <1L)
* Patients with deranged clotting profile (prothrombin time >3 seconds above control; activated partial thromboplastin time >10 seconds above control, platelet count <50000/µL)
* Patients already initiated on glucocorticoids
* Diagnosis of sarcoidosis possible on minimally invasive techniques such as skin biopsy or peripheral lymph node biopsy and failure to provide informed consent

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | 18 months
  The primary outcome is the diagnostic yield of the procedure defined as demonstration of granulomatous inflammation in two groups in patients finally labelled as sarcoidosis

SECONDARY OUTCOMES:
Safety | 18 months
  Occurrence of serious adverse events (pneumothorax, bleeding >100 ml, death) in the two groups
Diagnostic yield of individual sampling techniques | 18 months
  To study the diagnostic yield of EBUS-TBNA, conventional TBNA, TBLB and EBB

CONTACTS AND LOCATIONS:
Locations (1):
- Chest Clinic, PGIMER, Chandigarh, India

REFERENCES:
- [Derived] Gupta D, Dadhwal DS, Agarwal R, Gupta N, Bal A, Aggarwal AN. Endobronchial ultrasound-guided transbronchial needle aspiration vs conventional transbronchial needle aspiration in the diagnosis of sarcoidosis. Chest. 2014 Sep;146(3):547-556. doi: 10.1378/chest.13-2339. PMID 24481031